CLINICAL TRIAL: NCT06859151
Title: The Role of the Genital Tract Microbiota in Cervical Epithelial Cell DNA Methylation and the Increased Risk of Cervical Cancer Development
Brief Title: DNA Methylation and the Increased Risk of Cervical Cancer Development
Status: Not yet recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Muxuan Chen, Diagnostic Technician, Zhujiang Hospital
Other Study IDs: CALM2501
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer; Papillomavirus Infections
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biospecimen will include vaginal swabs, cervical exfoliated cells from reproductive tract of the volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control: HPV16(-) HPV18(-) TCT(-)
  Interventions: Other: Reproductive tract microbiota
- Case group 1: HPV16(+) /HPV18(+) TCT(-) CIN<2
  Interventions: Other: Reproductive tract microbiota
- Case group 2: HPV16(+) /HPV18(+) TCT(+) CIN<2
  Interventions: Other: Reproductive tract microbiota
- Case group 3: HPV16(+) /HPV18(+) TCT(+) CIN≥2+
  Interventions: Other: Reproductive tract microbiota

INTERVENTIONS:
Other: Reproductive tract microbiota — Reproductive tract microbiota

SUMMARY:
This study aims to investigate the correlation between reproductive tract microbiota and DNA methylation in cervical epithelial cells, as well as its impact on the development of cervical cancer, through a paired case-control clinical study

DETAILED DESCRIPTION:
This study is a multicenter matched case-control study. The inclusion and exclusion criteria are verified by collecting HPV test results, TCT examination results, and for the case group, participants' histopathological results are also collected. Participants who meet the inclusion and exclusion criteria have their HPV DNA test original secretion samples and TCT examination original cervical scrape cell samples (preserved in RNA preservative solution) collected. Enrollment involves dividing the samples into a discovery cohort of 800 cases and a validation cohort of 1200 cases. The discovery cohort undergoes multi-target DNA methylation testing, STDs pathogen testing, HPV E6/E7 testing, and metagenomic sequencing; the validation cohort undergoes PCR validation of DNA methylation sites related to cervical cancer, STDs pathogen testing, HPV E6/E7 testing, and metagenomic sequencing

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-50 years old, with a history of sexual activity
2. HPV and TCT tests are performed concurrently in the gynecology clinic
3. Those with abnormal HPV and TCT test results undergo tissue pathological testing

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Patients with immunological disorders or severe autoimmune diseases, such as AIDS, SLE
3. Those who have had organ transplants or are currently using immunosuppressive agents
4. Use of vaginal douching within 48 hours before sample collection
5. Use of vaginal probiotics within one month before sample collection
6. Use of vaginal antibiotics or antifungal treatments within one month before sample collection
7. History of surgery related to cervical intraepithelial neoplasia (CIN), including but not limited to conization of the cervix, LEEP procedures, etc.
8. Blood samples (avoid sampling during menstruation), insufficient remaining sample volume to support subsequent analysis needs, and samples not stored as required.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women aged 18 to 50
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in DNA methylation of cervical epithelial cells | Baseline (enrollment period)
  Changes in DNA methylation of cervical epithelial cells

SECONDARY OUTCOMES:
Cervical lesions (including different stages of development: normal, CIN 1, CIN 2, CIN 3, and cervical cancer), and sexually transmitted pathogens | Baseline (enrollment period)
  Cervical lesions (including different stages of development: normal, CIN 1, CIN 2, CIN 3, and cervical cancer), and sexually transmitted pathogens.

CONTACTS AND LOCATIONS:
Overall Officials: Muxuan Chen, Doctor, Principal Investigator — Department of Laboratory Medicine, Zhujiang Hospital, Southern Medical University